

Section of Surgical Oncology

# Feasibility Assessment of the Wake Forest Real-time Tracking System for Monitoring Patient Movement during Postoperative Recovery: Part 2

Informed Consent Form to Participate in Research Clancy J. Clark, Principal Investigator

#### INTRODUCTION

You are invited to be in a research study. Research studies are designed to gain scientific knowledge that may help other people in the future. You are being asked to take part in this study because you have recently undergone surgery. Your participation is voluntary. Please take your time in making your decision as to whether or not you wish to participate. Ask your study doctor or the study staff to explain any words or information contained in this informed consent document that you do not understand. You may also discuss the study with your friends and family.

#### WHY IS THIS STUDY BEING DONE?

The purpose of this research study is to study the use of a real-time tracking system called SPOT. The SPOT system is currently in use throughout the medical center to follow movement of important equipment, patients, and providers. Patients who are able to be physically active after surgery seem to have a better recovery. We would like to see if tracking patient movement with SPOT badges would be a good tool to measure physical activity after surgery.

# HOW MANY PEOPLE WILL TAKE PART IN THE STUDY?

Twenty (20) people will take part in this study.

#### WHAT IS INVOLVED IN THE STUDY?

If you take part in this study, we ask you questions or review your medical record for information about your medical condition, surgery, and physical function. The study team will have you walk in the hall during your recovery after surgery. You will be randomly assigned to walk in short intervals of a distance of 10 meters for a total of 40 meter OR to walk continuously for 40 meters.

During your walk, you will wear a small pedometer that measures the number of steps you are taking during your walk. The length, time, and distance of your walk will be determined by you. The study team will also evaluate your movement during your walk using the SPOT badge that


| | rage rors |
|-------------------------------|--------------------|
| | Adult Consent Forn |
| Version: | |
| IRB Template Version 06.15.17 | |



was provided at the time of your admission. Information regarding your physical activity and readiness for leaving the hospital will be collected by the study team.

#### HOW LONG WILL I BE IN THE STUDY?

You will be in the study for approximately one day after your surgery.

You can stop participating at any time. If you decide to stop participating in the study we encourage you to talk to the investigators or study staff first to learn about any potential health or safety consequences.

#### WHAT ARE THE RISKS OF THE STUDY?

The risk of harm or discomfort that may happen as a result of taking part in this research study is not expected to be more than in daily life or from routine physical or psychological examinations or tests. You should discuss the risk of being in this study with the study staff.

Taking part in this research study may involve providing information that you consider confidential or private. Efforts, such as coding research records, keeping research records secure and allowing only authorized people to have access to research records, will be made to keep your information safe.

#### ARE THERE BENEFITS TO TAKING PART IN THE STUDY?

If you agree to take part in this study, there may or may not be direct benefit to you. We hope the information learned from this study will benefit other people in the future. The benefits of participating in this study may be learning about your activity level while using the SPOT badge.

#### WHAT OTHER CHOICES ARE THERE?

This is not a treatment study. Your alternative is to not participate in this study.

# What About My Health Information?

In this research study, any new information we collect from you and/or information we get from your medical records about your health or behaviors is considered <u>Protected Health Information</u>.

We will make every effort to keep your Protected Health Information private. We will store records of your Protected Health Information in a cabinet in a locked office or on a password protected computer. Only the following people or organizations will be granted access to your Protected Health Information:

1) The study investigator and his/her staff, or others at Wake Forest University Health Sciences who oversee research


Adult Consent Form
Version:
IRB Template Version 06.15.17



2) Other people or laboratories providing services for this research project on behalf of Wake Forest University Health Sciences and Wake Forest University Baptist Medical Center

Some of the people, agencies and businesses that may receive and use your health information are the research sponsor; representatives of the sponsor assisting with the research; investigators at other sites who are assisting with the research; central laboratories, reading centers or analysis centers; the Institutional Review Board; representatives of Wake Forest University Health Sciences and North Carolina Baptist Hospital; representatives from government agencies such as the Food and Drug Administration (FDA) or the Office of Human Research Protections (OHRP), the Department of Health and Human Services (DHHS) and similar agencies in other countries.

Some of these people, agencies and businesses may further disclose your health information. If disclosed by them, your health information may no longer be covered by federal or state privacy regulations. Your health information may be disclosed if required by law. Your health information may be used to create information that does not directly identify you. This information may be used by other researchers. You will not be directly identified in any publication or presentation that may result from this study unless there are photographs or recorded media which are identifiable.

Any Protected Health Information collected from you in this study that is maintained in the research records will be kept for one year after the study is finished. At that time any research information not already in your medical record will either be destroyed or it will be de-identified.

You can tell Dr. Clancy J. Clark that you want to take away your permission to use and share your Protected Health Information at any time by sending a letter to this address:

Clancy J. Clark, MD
Department of General Surgery
Section of Surgical Oncology
Wake Forest University School of Medicine
Medical Center Blvd
Winston-Salem, NC 27157

However, if you take away permission to use your Protected Health Information you will not be able to be in the study any longer. We will stop collecting any more information about you, but any information we have already collected can still be used for the purposes of the research study.

By signing this form you give us permission to use your Protected Health Information for this study.

#### WHAT ARE THE COSTS?

Taking part in this study may lead to added costs to you or your insurance company. We will give you an estimate of what the added cost may be based on your particular situation and


Adult Consent Form

| Version: _ | | | |
|------------|--------|---------|----------|
| IRB Te | mplate | Version | 06.15.17 |



insurance coverage.

#### WILL YOU BE PAID FOR PARTICIPATING?

You will receive no payment or other compensation for taking part in this study.

#### WHO IS SPONSORING THIS STUDY?

This study is being sponsored by Wake Forest Baptist Health, Section on Surgical Oncology. The researchers do not, however, hold a direct financial interest in the sponsor or the product being studied.

# WHAT ARE MY RIGHTS AS A RESEARCH STUDY PARTICIPANT?

Taking part in this study is voluntary. You may choose not to take part or you may leave the study at any time. Refusing to participate or leaving the study will not result in any penalty or loss of benefits to which you are entitled. If you decide to stop participating in the study we encourage you to talk to the investigators or study staff first to learn about any potential health or safety consequences. The investigators also have the right to stop your participation in the study at any time. Examples of this could be because it is in your best medical interest, your condition worsened, new information becomes available, you had an unexpected reaction, you failed to follow instructions, or because the entire study has been stopped.

You will be given any new information we become aware of that would affect your willingness to continue to participate in the study.

## WHOM DO I CALL IF I HAVE QUESTIONS OR PROBLEMS?

For questions about the study or in the event of a research-related injury, contact the study investigator, Dr. Clancy J. Clark at 336-716-7207.

The Institutional Review Board (IRB) is a group of people who review the research to protect your rights. If you have a question about your rights as a research participant, or you would like to discuss problems or concerns, have questions or want to offer input, or you want to obtain additional information, you should contact the Chairman of the IRB at (336) 716-4542.

You will be given a copy of this signed consent form.

## **SIGNATURES**

I agree to take part in this study. I authorize the use and disclosure of my health information as described in this consent and authorization form. If I have not already received a copy of the Privacy Notice, I may request one or one will be made available to me. I have had a chance to ask questions about being in this study and have those questions answered. By signing this consent and authorization form, I am not releasing or agreeing to release the investigator, the sponsor, the institution or its agents from liability for negligence.

| | |
|-------------------------------|--------------------|
| | Adult Consent Form |
| Version: | |
| IRB Template Version 06.15.17 | |





| Subject Name (Printed): | | | |
|---------------------------|-------|-------------------|-------|
| Subject Signature: | Date: | Time: | am pm |
| Person Obtaining Consent: | Date: | Time <sup>.</sup> | am pn |


Adult Consent Form

Version: \_\_\_\_\_\_ IRB Template Version 06.15.17